CLINICAL TRIAL: NCT04147273
Title: Determination of Postprandial Glycemic Responses by Continuous Glucose Monitoring in a Real-World Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West German Center of Diabetes and Health (Other)
Collaborators: Bionorica SE (Industry)
Responsible Party: Principal Investigator, Stephan Martin, Director of the West German Center of Diabetes and Health, Head of Diabetology, West German Center of Diabetes and Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 11
Record Dates: First submitted 2019-06-24; First posted 2019-11-01 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Postprandial Glucose Response; Glycaemic Index; Continous Glucose Measurement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation of CGM compared with standard measurements (Other): Two products were studied: white bread (Butter Toast®, Golden Toast, Wittenberg, Germany) and whole grain bread (1688 Mehrkorn®, Harry-Brot, Schenefeld, Germany). One portion (containing 50 g digestible carbohydrates) was eaten immediately before the beginning of the test in the morning after an overnight fast of at least 10 h. Before testing, participants ate as usual on the previous day without a standard meal and refrained from consuming alcohol and exercising for 72 h. A 200-ml glucose drink (Accu-Chek Dextrose O.G.-T. Saft®, Roche Diabetes Care, Mannheim, Germany), containing also 50 g of carbohydrates, was used as the reference product.
  Interventions: Device: Determination of postprandial glucose response by continuous glucose measurement after consuming different carbohydrate containing foods

INTERVENTIONS:
Device: Determination of postprandial glucose response by continuous glucose measurement after consuming different carbohydrate containing foods — One day prior to the study beginning, participants were equipped with a CGM system (FreeStyle Libre®, Abbott Diabetes Care, Alameda, CA, USA). This CGM system provides glucose recordings every 15 min over a period of 14 days. The glucose data were downloaded manually by a scan with a handheld device.
  On the second day of the study, participants consumed portions of these three test products containing 50 g of available carbohydrate on 3 separate days without a washout period. The products were tested in random order at the same time of the morning after a 10 h overnight fast. Venous blood samples were collected at 0, 15, 30, 45, 60, 75, 90, 105 and 120 min postprandial by inserting an intravenous cannula into a forearm vein. Capillary blood samples were obtained through finger pricking. Blood glucose levels in these samples were measured with a high quality SMBG system (ContourXT/Contour next, Ascensia Diabetes Care, Leverkusen, Deutschland, Germany).

SUMMARY:
Self-monitoring of blood glucose using capillary glucose testing has a number of shortcomings compared to continuous glucose monitoring (CGM). We aimed to compare these two methods and used blood glucose measurements in venous blood as a reference. Despite considerable inter-individual variability of postprandial glycemic responses, CGM evaluated postprandial glycemic excursions which had comparable results compared to standard blood glucose measurements under real-life conditions.

DETAILED DESCRIPTION:
Self-monitoring of blood glucose using capillary glucose testing (C) has a number of shortcomings compared to continuous glucose monitoring (CGM). We aimed to compare these two methods and used blood glucose measurements in venous blood (IV) as a reference. Postprandial blood glucose levels were measured after 50 g oral glucose load and after the consumption of a portion of different foods containing 50 g of carbohydrates. We also evaluated the associations between postprandial glucose responses and the clinical characteristics of the participants at the beginning of the study. Incremental area under the curve (AUCi) of postprandial blood glucose was calculated for 1 h (AUCi 0-60) and 2 h (AUCi 0-120). Despite considerable inter-individual variability of postprandial glycemic responses, CGM evaluated postprandial glycemic excursions which had comparable results compared to standard blood glucose measurements under real-life conditions.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old

Exclusion Criteria:

* acute diseases, severe illness with in-patient treatment during the last 3 months, weight change >2 kg/week during the last month, smoking secession during the last 3 months, drugs for active weight reduction, chronic medication

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Postprandial glucose response | 1 and 2 hours after food consumption
  postprandial glycemic changes after consuming different carbohydrate containing foods

SECONDARY OUTCOMES:
incremental AUC (AUCi) of postprandial glucose excursions | 1 and 2 hours after food consumption
  after consuming different carbohydrate containing foods

CONTACTS AND LOCATIONS:
Locations (1):
- West-German Center of Diabetes and Health, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: No